CLINICAL TRIAL: NCT02418078
Title: Retrospective Analysis of the Geriatric Patients Underwent Unilateral Inguinal Herniorrhaphy at Our Institution
Brief Title: Retrospective Analysis of the Geriatric Patients Underwent Unilateral Inguinal Herniorrhaphy
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, DR, Diskapi Teaching and Research Hospital
Other Study IDs: Geriatri Hernia
Record Dates: First submitted 2015-02-14; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-02

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthesia, Local

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Geriatri: patients ageing ≥ 65 yr undergoing herniorrhaphy with local infiltration anesthesia and sedation
  Interventions: Procedure: local infiltration anesthesia and sedation
- non-geriatri: patients ageing 19-64 yr undergoing herniorrhaphy with local infiltration anesthesia and sedation
  Interventions: Procedure: local infiltration anesthesia and sedation

INTERVENTIONS:
Procedure: local infiltration anesthesia and sedation — the surgical site is infiltrated with local anesthetic agents and the patients are sedated with intravenous agents
  Other Names: local anesthesia and sedation

SUMMARY:
The aim of this study is to compare the geriatric patients with the non-geriatrics undergoing outpatient unilateral herniorrhapy in terms of local anesthesia, sedation, recovery and early morbidity.

DETAILED DESCRIPTION:
A retrospective data analysis will be conducted and the patient records will be evaluated for patient characteristics local anesthesia, sedation, recovery and early morbidity.

ELIGIBILITY:
Inclusion Criteria:

patients with a unilateral inguinal hernia undergoing herniorrhaphy

Exclusion Criteria:

none

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a unilateral inguinal hernia
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
discharge time | postoperative 2 hours
discharge delay | postoperative 2 hours
local anesthetic doses | intraoperative
sedative doses | intraoperative

SECONDARY OUTCOMES:
complications (hypertension, tachycardia, bradycardia, hypotension, nausea, vomiting) | intraoperative
early morbidity | postoperative 2 hours
morbidity | postopative 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Kulacoglu, Prof, Study Director — Diskapi Teaching and Research Hospital
Locations (1):
- Dıskapı TRH, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Mattila K, Hynynen M; Intensium Consortium Study Group. Day surgery in Finland: a prospective cohort study of 14 day-surgery units. Acta Anaesthesiol Scand. 2009 Apr;53(4):455-63. doi: 10.1111/j.1399-6576.2008.01895.x. Epub 2009 Feb 23. PMID 19239413
- [Result] Majholm B, Engbaek J, Bartholdy J, Oerding H, Ahlburg P, Ulrik AM, Bill L, Langfrits CS, Moller AM. Is day surgery safe? A Danish multicentre study of morbidity after 57,709 day surgery procedures. Acta Anaesthesiol Scand. 2012 Mar;56(3):323-31. doi: 10.1111/j.1399-6576.2011.02631.x. PMID 22335277
- [Result] Dallas KB, Froylich D, Choi JJ, Rosa JH, Lo C, Colon MJ, Telem DA, Divino CM. Laparoscopic versus open inguinal hernia repair in octogenarians: a follow-up study. Geriatr Gerontol Int. 2013 Apr;13(2):329-33. doi: 10.1111/j.1447-0594.2012.00902.x. Epub 2012 Jun 21. PMID 22726915